CLINICAL TRIAL: NCT03345095
Title: A Phase III Trial of Marizomib in Combination With Standard Temozolomide-based Radiochemotherapy Versus Standard Temozolomide-based Radiochemotherapy Alone in Patients With Newly Diagnosed Glioblastoma
Brief Title: A Phase III Trial of With Marizomib in Patients With Newly Diagnosed Glioblastoma
Acronym: MIRAGE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Collaborators: Celgene (Industry); Canadian Cancer Trials Group (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EORTC-BTG-1709
Record Dates: First submitted 2017-11-07; First posted 2017-11-17 (Actual); Results first posted 2024-01-31 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Newly Diagnosed Glioblastoma
Keywords: Marizomib; Temozolomide; Glioblastoma; Phase III
MeSH Terms: conditions — Glioblastoma | interventions — marizomib; Temozolomide; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Experimental Arm (Experimental): Radiotherapy + Temozolomide + Marizomib followed by adjuvant Temozolomide + Marizomib
  Interventions: Drug: Marizomib; Drug: Temozolomide; Radiation: radiotherapy
- Standard Arm (Active Comparator): Radiotherapy + Temozolomide followed by adjuvant Temozolomide
  Interventions: Drug: Temozolomide; Radiation: radiotherapy

INTERVENTIONS:
Drug: Marizomib — Intravenous administration of Marizomib
  Arms: Experimental Arm
Drug: Temozolomide — Oral Administration of Temozolomide
  Other Names: TMZ
Radiation: radiotherapy — 60 Gy in 30 fractions over 6 weeks
  Other Names: RT

SUMMARY:
The standard of care for newly diagnosed glioblastoma includes surgery, involved-field radiotherapy, and concomitant and six cycles of maintenance temozolomide chemotherapy, however the prognosis remains dismal. Marizomib has been tested in patients with newly diagnosed and recurrent glioblastoma in phase I and phase II studies. In patients with recurrent glioblastoma, marizomib was administered as a single agent or in combination with bevacizumab (NCT02330562). Based on encouraging observations, a phase I/II trial of marizomib in combination with Temozolomide+Radiotherapy(TMZ/RT) followed by Temozolomide (TMZ) in newly diagnosed glioblastoma has been launched (NCT02903069) which explores safety and tolerability of this triple combination and which shall help to determine the dose for further clinical trials in glioblastoma. In this context, given that marizomib has been established as a safe addition to the standard TMZ/RT -->TMZ, a phase III study is considered essential to establishing its impact on overall survival.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed newly diagnosed glioblastoma (WHO grade IV)
* Tumor resection (gross total or partial), or biopsy only
* Availability of formalin-fixed paraffin-embedded (FFPE) tumor block or 24 unstained slides for o6-methylguanine-DNA-methyltransferase (MGMT) analysis
* Patient must be eligible for standard TMZ/RT + TMZ
* Karnofsky performance score (KPS) ≥ 70
* Recovered from effects of surgery, postoperative infection and other complications of surgery (if any)
* The patient is at least 18 years of age on day of signing informed consent
* Stable or decreasing dose of steroids for at least 1 week prior to inclusion
* The patient has a life expectancy of at least 3 months
* Patient has undergone a brain MRI within 14 days of randomization but after intervention (resection or biopsy)
* The patient shows adequate organ functions as assessed by the specified laboratory values within 2 weeks prior to randomization defined as adequate bone marrow, renal and hepatic function within the following ranges:

  * white blood cell count (WBC) ≥ 3×10*9/L
  * absolute neutrophil count (ANC) ≥ 1.5×10*9/L
  * Platelet count of ≥ 100×10*9/L independent of transfusion
  * Hemoglobin ≥ 10 g/dl
  * Total Bilirubin ≤ 1.5 upper limit of normal (ULN)
  * Alanine aminotransferase (ALT), aspartate aminotransferase (AST), alkaline phosphatase (ALP) ≤ 2.5 × ULN
  * Serum creatinine < 1.5 x ULN or creatinine clearance (CrCl) > 30 mL/min(using the Cockcroft-Gault formula)
* Women of child bearing potential (WOCBP) must have a negative urine or serum pregnancy test within 7 days prior to the first dose of study treatment.
* Patients of childbearing / reproductive potential must agree to use adequate birth control measures, as defined by the investigator, during the study treatment period and for at least 6 months after the last study treatment. A highly effective method of birth control is defined as those which result in low failure rate (i.e. less than 1 percent per year) when used consistently and correctly. Patients must also agree not to donate sperm during the study and for 6 months after receiving the last dose of study treatment.
* Women who are breast feeding must agree to discontinue nursing prior to the first dose of study treatment and until 6 months after the last study treatment.
* Ability to take oral medication
* Ability to understand the requirements of the study, provide written informed consent and authorization of use and disclosure of protected health information, and agree to abide by the study restrictions and return for the required assessments.
* Before patient registration/randomization, written informed consent must be given according to International Council for Harmonisation (ICH) / Good clinical practice (GCP), and national/local regulations.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 749 (Actual)
Dates: Start 2018-07-26 (Actual); Primary Completion 2022-08-23 (Actual); Study Completion 2023-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Roth, Principal Investigator — EORTC Study Coordinator
Locations (82):
- United States (9):
  - Mayo Clinic Scottsdale, Scottsdale, Arizona
  - University of California at Irvine, Orange, California
  - University of California, San Francisco, California
  - John Wayne Cancer Institute, Santa Monica, California
  - University of Florida, Gainesville, Florida
  - Mayo Clinic, Jacksonville, Florida
  - Mayo Clinic, Rochester, Minnesota
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Penn State College of Medicine, Hershey Medical Center-Penn State Neuroscience Institute, Hershey, Pennsylvania
- Austria (3):
  - Innsbruck Universitaetsklinik, Innsbruck
  - Kepler University Hospital, Linz
  - Medical University Vienna - General Hospital AKH, Vienna
- Belgium (7):
  - Onze Lieve Vrouw Ziekenhuis, Aalst
  - GasthuisZusters Antwerpen - Sint-Augustinus, Antwerp
  - Hopitaux Universitaires Bordet-Erasme - Hopital Universitaire Erasme, Brussels
  - Cliniques Universitaires Saint-Luc, Brussels
  - Grand Hopital de Charleroi - Grand Hôpital de Charleroi - Site Notre Dame, Charleroi
  - Universitair Ziekenhuis Gent, Ghent
  - C.H.U. Sart-Tilman, Liège
- Canada (23):
  - Saint John Regional Hospital, Saint John, New Brunswick
  - London Regional Cancer Center, London, Ontario
  - Ottawa Health Research Institute, Ottawa, Ontario
  - Windsor Regional Cancer Centre, Windsor, Ontario
  - Centre Hospitalier Universitaire de Sherbrooke-Fleurimont, Sherbrooke, Quebec
  - BCCA - Abbotsford Centre, Abbotsford
  - Tom Baker Cancer Centre, Calgary
  - Regional Cancer Program of Hopital Reg. de Sudbury Reg. Hospital, Greater Sudbury
  - QEII Health Sciences Centre-Capital District Health Authority, Halifax
  - Hamilton Health Sciences, Juravinski Cancer Centre, Hamilton
  - Kingston Health Sciences Centre, Kingston
  - Montreal Neurological Institute and Hospital McGill University, Montreal
  - CHUM - Centre Hospitalier de l'Université de Montreal - Hopital Notre-Dame, Montreal
  - Hopital Du Sacre-Coeur De Montreal, Montreal
  - CHU de Quebec-Hopital l'Enfant-Jesus (HEJ), Québec
  - Allan Blair Cancer Centre, Regina
  - Sault Area Hospital, Sault Ste. Marie
  - Odette Cancer Centre - Sunnybrook Health Sciences Centre, Toronto
  - University Health Network - Oci / Princess Margaret Hospital, Toronto
  - Centre hospitalier regional de Trois-Rivieres, Trois-Rivières
  - BC Cancer Agency, Vancouver
  - Bcca - Vancouver Island Cancer Centre, Victoria
  - Cancercare Manitoba, Winnipeg
- Denmark (2):
  - Aarhus University Hospitals - Aarhus University Hospital, Aarhus
  - University Hospitals Copenhagen - Rigshospitalet, Copenhagen
- France (6):
  - Centre Hospitalier Departemental Vendée, La Roche-sur-Yon, Vendee
  - CHU de Lyon - CHU Lyon - Hopital neurologique Pierre Wertheimer, Bron
  - CHRU de Lille, Lille
  - Institut de Cancerologie de l'Ouest, Nantes
  - Assistance Publique - Hopitaux de Paris - La Pitie Salpetriere, Paris
  - Gustave Roussy, Villejuif
- Germany (10):
  - Universitaetsklinikum Bonn, Bonn
  - Universitaetsklinik Erlangen-Neurologische Klinik, Erlangen
  - Klinikum Der J.W. Goethe Universitaet-Klinik und Poliklinik fur Neurochirurgie, Frankfurt
  - UniversitaetsKlinikum Heidelberg - Head Hospital, Heidelberg
  - Universitaetsklinikum Leipzig-Klinik für Strahlentherapie und Radioonkologie, Leipzig
  - Johannes Gutenberg Universitaetskliniken - Mainz University Medical Center, Mainz
  - UniversitaetsMedizin Mannheim, Mannheim
  - Technische Universitaet Muenchen - Klinikum Rechts Der Isar, München
  - Universitaetskliniken Regensburg, Regensburg
  - Universitaetsklinikum Tuebingen- Crona Kliniken, Tübingen
- Netherlands (9):
  - Catharina Ziekenhuis, Eindhoven, North Brabant
  - Spaarne Gasthuis - Vrije Universiteit Medisch Centrum, Amsterdam
  - The Netherlands Cancer Institute-Antoni Van Leeuwenhoekziekenhuis, Amsterdam
  - University Medical Center Groningen, Groningen
  - Academisch Ziekenhuis Maastricht, Maastricht
  - Radboud University Medical Center Nijmegen, Nijmegen
  - Erasmus MC, Rotterdam
  - Medisch Centrum Haaglanden - Westeinde, The Hague
  - Universitair Medisch Centrum - Academisch Ziekenhuis, Utrecht
- Oslo University Hospital - Radiumhospitalet, Oslo, Norway
- Spain (5):
  - Institut Catala d'Oncologia - ICO Badalona - Hospital Germans Trias i Pujol (Institut Catala D'Oncologia), Badalona
  - Hospital Clinic Universitari de Barcelona, Barcelona
  - Institut Catala D'Oncologia, L'Hospitalet de Llobregat
  - Hospital Universitario 12 De Octubre, Madrid
  - Clinica Universidad de Navarra - Clinica Universitaria De Navarra, Pamplona
- Switzerland (4):
  - University Hospital of Geneva, Geneva
  - Centre Hospitalier Universitaire Vaudois, Lausanne
  - Kantonsspital, Sankt Gallen
  - UniversitaetsSpital, Zurich
- United Kingdom (3):
  - NHS Lothian - Western General Hospital, Edinburgh
  - Guy's and St Thomas' NHS - Guy s and St Thomas' NHS - Guy's Hospital, London
  - Sheffield Teaching Hospitals NHS Foundation Trust - Weston Park Hospital, Sheffield

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patient registration was accepted from authorized investigators. Patients were registered on the Electronic Data Capture system. To access it, the investigator needed a user name and a password which were provided by the EORTC Headquarters. In case of problems investigators could contact the EORTC Clinical Data Manager. A Subject Identifier was allocated to the patient. This number allowed the identification of the patient in the Electronic Data Capture.
Pre-assignment Details: Eligibility criteria were checked at time of randomization. Once eligibility had been verified, treatment was randomly allocated to the patient, together with a sequential patient identification number. This number allowed the identification of the patients in the Electronic Data Capture system that was used to complete the Case Report Forms.
Period: Overall Study
Arm/Group | Experimental Arm | Standard Arm
Started | 374 | 375
Completed | 125 | 8
Not Completed | 249 | 367
Not completed — Lack of Efficacy | 184 | 156
Not completed — Adverse Event | 36 | 118
Not completed — Withdrawal by Subject | 22 | 59
Not completed — Physician Decision | 3 | 18
Not completed — Death | 2 | 4
Not completed — Other reasons | 2 | 11
Not completed — Protocol Violation | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Experimental Arm | Standard Arm | Total
Number analyzed (Participants) | 374 | 375 | 749
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 287 | 276 | 563
  >=65 years | 87 | 99 | 186
Age, Continuous [Median (Full Range); unit: years] | 58.5 [21 to 79] | 58.0 [20 to 79] | 58.0 [20 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 119 | 142 | 261
  Male | 255 | 233 | 488
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 7 | 5 | 12
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 2 | 0 | 2
  White | 279 | 290 | 569
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 85 | 79 | 164
Region of Enrollment [Number; unit: participants]
  Canada | 104 | 108 | 212
  Austria | 6 | 7 | 13
  Netherlands | 45 | 44 | 89
  Belgium | 30 | 32 | 62
  United States | 21 | 19 | 40
  Norway | 4 | 4 | 8
  Denmark | 9 | 10 | 19
  United Kingdom | 8 | 7 | 15
  France | 55 | 54 | 109
  Switzerland | 20 | 24 | 44
  Germany | 38 | 37 | 75
  Spain | 34 | 29 | 63
Karnofsky Performance Status [Count of Participants; unit: Participants] — The Karnofsky Performance Status Index allows patients to be classified as to their functional impairment. This can be used to compare effectiveness of different therapies and to assess the prognosis in individual patients. The lower the Karnofsky score, the worse the survival for most serious illnesses. 100 Normal no complaints; no evidence of disease. 90 Able to carry on normal activity; minor signs or symptoms of disease. 80 Normal activity with effort; some signs or symptoms of disease. 70 Cares for self; unable to carry on normal activity or to do active work.
  Participants
    70/80 | 126 | 123 | 249
    90/100 | 248 | 252 | 500
Extent of surgery [Count of Participants; unit: Participants]
  Gross total | 192 | 192 | 384
  Partial/biopsy | 182 | 183 | 365

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS)
Description: Overall Survival (OS): OS is defined as the number of days from date of randomization to the date of death due to any cause. If a patient has not died, the data will be censored at the last date documented to be alive.
Time Frame: From the date of randomization up to the date of death, assessed up to 49 months
Population: Analysis population is Intention-to-treat population (ITT): All randomized patients will be analyzed in the arm they were allocated by randomization
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Experimental Arm | Standard Arm
Number analyzed (Participants) | 309 | 307
Months | 16.13 [14.92 to 17.77] | 15.08 [13.73 to 16.99]

2. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS is defined as the number of days from date of randomization to the date of earliest disease progression based on Response Assessment in Neuro-Oncology criteria (by investigator) or to the date of death due to any cause, if disease progression does not occur. Patients for whom neither death nor progression have been documented were censored on the date of the last radiological assessment that the patient was progression-free. If a patient with no post-baseline radiological assessment then the data were censored at the date of randomization. Patients with two or more missing response assessments prior to a visit with documented disease progression (or death) were censored at the last visit where the patient was documented to be progression free. Patients who received new anti-cancer therapy or cancer-related surgery prior to progression or death were not censored at the last assessment where the patient was documented as progression free prior to the new therapy.
Time Frame: From the date of randomization until the date of first objective progression or the date of patient's death whichever occurs first, assessed up to 49 months
Population: The analysis population is Intention-to-treat population (ITT): All randomized patients will be analyzed in the arm they were allocated by randomization.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Experimental Arm | Standard Arm
Number analyzed (Participants) | 309 | 307
Months | 6.34 [5.82 to 7.85] | 6.11 [4.93 to 7.29]

3. Secondary Outcome: Health-related Quality of Life (HRQol)
Description: HRQoL was assessed with the EORTC Quality of Life Questionnaire (QLQ-C30) version 3. The primary HRQol score is Physical Functioning. It is reported at week 16 during the Temozolomide (TMZ) maintenance phase. Physical functioning score is ranging 0 to 100. A large scores indicate a good physical functioning. A negative difference indicates a worsening physical functioning.
Time Frame: From randomization until progression or death which ever occurs first, reported at week 16 by the mean difference from baseline assessment.
Population: At week 16 during the TMZ maintenance phase, HRQol was obtained from 212 patients in the Experimental arm and 207 patients in the Standard arm.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Experimental Arm | Standard Arm
Number analyzed (Participants) | 212 | 207
score on a scale | -11.8 [-15.0 to -8.7] | -5.4 [-8.0 to -2.9]
Statistical Analysis 1: Comparison: Experimental Arm vs Standard Arm; Test type: Superiority; p = 0.0004, Wilcoxon (Mann-Whitney); Mean Difference (Net) = -6.4, 95% CI 2-sided [-8.6 to -2.5]

4. Secondary Outcome: Mini Mental State Examination (MMSE)
Description: MMSE is a brief, standardized tool to grade patients' neurocognitive function. It is an 11-question measure that tests five areas of neurocognitive function: orientation, registration, attention and calculation, recall, and language. A large MMSE score indicates a good cognitive functioning. The maximum MMSE score is 30 which corresponds to the best neurocognitive function and minimum MMSE score is 0 the worst neurocognitive function.The patient's neurocognitive function are considered 'impaired' if MMSE is 26 or less and 'normal' if it is 27 or more. MMSE has been validated and extensively used in both clinical practice and research. It is reported at week 16 during the Temozolomide (TMZ) maintenance phase. A negative difference indicates a worsening cognitive functioning. Difference range reported in the data table is min -19 and max 10. The mean difference is reported with 95% confidence interval (CI). A CI which excludes 0 indicates a significant mean MMSE score change.
Time Frame: From the date of randomization until end of treatment. It is reported at week 16 by the mean difference from baseline assessment.
Population: At week 16 during the TMZ maintenance phase, HRQol was obtained from 180 patients in the Experimental arm and 166 patients in the Standard arm.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Experimental Arm | Standard Arm
Number analyzed (Participants) | 180 | 166
score on a scale | -0.95 [-1.51 to -0.38] | -0.39 [-0.82 to 0.04]
Statistical Analysis 1: Comparison: Experimental Arm vs Standard Arm; Test type: Superiority; p = 0.15, Wilcoxon (Mann-Whitney); Mean Difference (Net) = -0.55, 95% CI 2-sided [-1.27 to 0.16]

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) were collected from first dose of radiotherapy up to 49 months after patient enrolment in the study. All-Cause Mortality was assessed through study completion, up to 49 months after patient enrolment in the study.
Description: Both serious and non-serious AEs were collected. We reported serious adverse events (SAEs) and all AEs. Non serious AEs are accounted for in the all AEs report. All AEs report is included in the Other (Not Including Serious) section. All-cause mortality was assessed in the intent to treat population defined as all randomized patients. SAEs and all AEs were assessed in the randomized patients who have started their allocated treatments
Arm/Group | Experimental Arm | Standard Arm
All-Cause Mortality (participants affected / at risk) | 55/309 | 57/307
Serious Adverse Events (participants affected / at risk) | 114/305 | 80/297
Other Adverse Events (participants affected / at risk) | 300/305 | 283/297
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Experimental Arm (N=305) | Standard Arm (N=297)
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Febrile Neutropenia (Blood and lymphatic system disorders) | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 2 | 1
Neutropenia (Blood and lymphatic system disorders) | 3 | 1
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 7 | 1
Angina Pectoris (Cardiac disorders) | 1 | 0
Atrial Flutter (Cardiac disorders) | 1 | 0
Diplopia (Ear and labyrinth disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 1
Enterocolitis (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0
Gastrointestinal Inflammation (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 7 | 1
Upper Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 5 | 2
Catheter Site Thrombosis (General disorders) | 1 | 0
Fatigue (General disorders) | 4 | 0
Gait Disturbance (General disorders) | 1 | 2
General Physical Health Deterioration (General disorders) | 4 | 5
Impaired Healing (General disorders) | 0 | 1
Influenza Like Illness (General disorders) | 0 | 1
Oedema Peripheral (General disorders) | 0 | 1
Peripheral Swelling (General disorders) | 1 | 0
Pyrexia (General disorders) | 2 | 3
Vascular Device Occlusion (General disorders) | 1 | 0
Drug-Induced Liver Injury (Hepatobiliary disorders) | 1 | 0
Anal Abscess (Infections and infestations) | 1 | 0
Bacterial Infection (Infections and infestations) | 0 | 1
Brain Abscess (Infections and infestations) | 0 | 1
Covid-19 (Infections and infestations) | 0 | 1
Cystitis (Infections and infestations) | 2 | 1
Cytomegalovirus Infection (Infections and infestations) | 0 | 1
Device Related Infection (Infections and infestations) | 1 | 0
Device Related Sepsis (Infections and infestations) | 1 | 0
Enterocolitis Infectious (Infections and infestations) | 1 | 0
Gastroenteritis Viral (Infections and infestations) | 1 | 0
Herpes Zoster Infection Neurological (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 0 | 1
Lower Respiratory Tract Infection (Infections and infestations) | 1 | 0
Meningitis Bacterial (Infections and infestations) | 1 | 1
Pneumocystis Jirovecii Pneumonia (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 5 | 1
Pneumonia Chlamydial (Infections and infestations) | 1 | 0
Retinitis (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 2 | 0
Septic Shock (Infections and infestations) | 1 | 0
Staphylococcal Bacteraemia (Infections and infestations) | 1 | 0
Subdural Abscess (Infections and infestations) | 1 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 1 | 0
Urinary Tract Infection (Infections and infestations) | 1 | 1
Urosepsis (Infections and infestations) | 1 | 0
Viral Rash (Infections and infestations) | 0 | 1
Wound Infection (Infections and infestations) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 5 | 1
Femoral Neck Fracture (Injury, poisoning and procedural complications) | 0 | 1
Head Injury (Injury, poisoning and procedural complications) | 1 | 0
Pneumocephalus (Injury, poisoning and procedural complications) | 0 | 1
Pseudomeningocele (Injury, poisoning and procedural complications) | 0 | 1
Radiation Necrosis (Injury, poisoning and procedural complications) | 1 | 0
Radius Fracture (Injury, poisoning and procedural complications) | 0 | 1
Spinal Fracture (Injury, poisoning and procedural complications) | 1 | 0
Subdural Haematoma (Injury, poisoning and procedural complications) | 0 | 1
Tendon Rupture (Injury, poisoning and procedural complications) | 1 | 0
Alanine Aminotransferase Increased (Investigations) | 1 | 0
Aspartate Aminotransferase Increased (Investigations) | 1 | 0
Blood Creatinine Increased (Investigations) | 1 | 1
Lymphocyte Count Decreased (Investigations) | 1 | 0
Neutrophil Count Decreased (Investigations) | 1 | 1
Platelet Count Decreased (Investigations) | 2 | 7
White Blood Cell Count Decreased (Investigations) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1
Steroid Diabetes (Metabolism and nutrition disorders) | 0 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 1 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Brain Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Glioblastoma Multiforme (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant Neoplasm Progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8 | 5
Metastases To Meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Neoplasm Progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Peritumoural Oedema (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Squamous Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Akathisia (Nervous system disorders) | 1 | 0
Aphasia (Nervous system disorders) | 2 | 1
Ataxia (Nervous system disorders) | 4 | 0
Balance Disorder (Nervous system disorders) | 1 | 0
Brain Oedema (Nervous system disorders) | 8 | 8
Brain Stem Haematoma (Nervous system disorders) | 1 | 0
Cerebral Haemorrhage (Nervous system disorders) | 2 | 0
Cerebral Ischaemia (Nervous system disorders) | 1 | 0
Cerebral Venous Thrombosis (Nervous system disorders) | 1 | 0
Clonus (Nervous system disorders) | 0 | 1
Cognitive Disorder (Nervous system disorders) | 1 | 0
Coordination Abnormal (Nervous system disorders) | 1 | 0
Depressed Level Of Consciousness (Nervous system disorders) | 3 | 0
Dizziness (Nervous system disorders) | 1 | 1
Dysarthria (Nervous system disorders) | 1 | 0
Encephalopathy (Nervous system disorders) | 1 | 1
Epilepsy (Nervous system disorders) | 4 | 3
Generalised Tonic-Clonic Seizure (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 6 | 2
Hemiparesis (Nervous system disorders) | 3 | 2
Hydrocephalus (Nervous system disorders) | 2 | 2
Intracranial Pressure Increased (Nervous system disorders) | 2 | 0
Ischaemic Stroke (Nervous system disorders) | 1 | 0
Lethargy (Nervous system disorders) | 1 | 0
Leukoencephalopathy (Nervous system disorders) | 1 | 0
Motor Dysfunction (Nervous system disorders) | 2 | 1
Nervous System Disorder (Nervous system disorders) | 2 | 1
Neurological Decompensation (Nervous system disorders) | 4 | 1
Neurological Symptom (Nervous system disorders) | 1 | 0
Neuromyelitis Optica Spectrum Disorder (Nervous system disorders) | 1 | 0
Nystagmus (Nervous system disorders) | 2 | 0
Partial Seizures (Nervous system disorders) | 1 | 0
Post Herpetic Neuralgia (Nervous system disorders) | 1 | 0
Pyramidal Tract Syndrome (Nervous system disorders) | 0 | 1
Radicular Pain (Nervous system disorders) | 1 | 0
Seizure (Nervous system disorders) | 15 | 14
Somnolence (Nervous system disorders) | 0 | 1
Status Epilepticus (Nervous system disorders) | 1 | 1
Subdural Effusion (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 0 | 3
Vasogenic Cerebral Oedema (Nervous system disorders) | 3 | 3
Agitation (Psychiatric disorders) | 3 | 0
Anxiety (Psychiatric disorders) | 1 | 0
Confusional State (Psychiatric disorders) | 7 | 3
Delirium (Psychiatric disorders) | 4 | 2
Delusion (Psychiatric disorders) | 1 | 0
Hallucination (Psychiatric disorders) | 7 | 0
Hallucination, Visual (Psychiatric disorders) | 2 | 1
Impulsive Behaviour (Psychiatric disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 1 | 0
Irritability (Psychiatric disorders) | 2 | 0
Mania (Psychiatric disorders) | 1 | 0
Paranoia (Psychiatric disorders) | 1 | 0
Psychomotor Retardation (Psychiatric disorders) | 1 | 0
Psychotic Disorder (Psychiatric disorders) | 1 | 0
Acute Kidney Injury (Renal and urinary disorders) | 1 | 0
Renal Failure (Renal and urinary disorders) | 1 | 0
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 1 | 0
Stevens-Johnson Syndrome (Skin and subcutaneous tissue disorders) | 1 | 0
Deep Vein Thrombosis (Vascular disorders) | 2 | 0
Embolism (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 0
Jugular Vein Thrombosis (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Experimental Arm (N=305) | Standard Arm (N=297)
Anaemia (Blood and lymphatic system disorders) | 16 | 18
Febrile Neutropenia (Blood and lymphatic system disorders) | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 8 | 6
Lymphopenia (Blood and lymphatic system disorders) | 18 | 18
Neutropenia (Blood and lymphatic system disorders) | 13 | 11
Pancytopenia (Blood and lymphatic system disorders) | 2 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 27 | 29
Angina Pectoris (Cardiac disorders) | 1 | 0
Atrial Fibrillation (Cardiac disorders) | 1 | 1
Atrial Flutter (Cardiac disorders) | 1 | 0
Cardiac Failure (Cardiac disorders) | 1 | 0
Palpitations (Cardiac disorders) | 5 | 2
Sinus Bradycardia (Cardiac disorders) | 0 | 1
Sinus Tachycardia (Cardiac disorders) | 2 | 2
Supraventricular Tachycardia (Cardiac disorders) | 0 | 1
Tachycardia (Cardiac disorders) | 2 | 1
Deafness (Ear and labyrinth disorders) | 0 | 3
Ear Congestion (Ear and labyrinth disorders) | 1 | 0
Ear Discomfort (Ear and labyrinth disorders) | 4 | 1
Ear Pain (Ear and labyrinth disorders) | 5 | 3
Hyperacusis (Ear and labyrinth disorders) | 1 | 1
Hypoacusis (Ear and labyrinth disorders) | 7 | 0
Presbyacusis (Ear and labyrinth disorders) | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 11 | 5
Vertigo (Ear and labyrinth disorders) | 25 | 3
Vestibular Disorder (Ear and labyrinth disorders) | 2 | 0
Cushing's Syndrome (Endocrine disorders) | 1 | 0
Cushingoid (Endocrine disorders) | 7 | 5
Altered Visual Depth Perception (Eye disorders) | 1 | 0
Asthenopia (Eye disorders) | 1 | 1
Blindness (Eye disorders) | 1 | 0
Cataract (Eye disorders) | 1 | 2
Diplopia (Eye disorders) | 22 | 2
Dry Eye (Eye disorders) | 4 | 1
Dyschromatopsia (Eye disorders) | 1 | 0
Eye Discharge (Eye disorders) | 1 | 0
Eye Inflammation (Eye disorders) | 0 | 1
Eye Irritation (Eye disorders) | 2 | 0
Eye Pain (Eye disorders) | 2 | 3
Eye Paraesthesia (Eye disorders) | 0 | 1
Eyelid Function Disorder (Eye disorders) | 0 | 1
Eyelid Oedema (Eye disorders) | 1 | 0
Eyelid Ptosis (Eye disorders) | 1 | 0
Glare (Eye disorders) | 1 | 0
Hypermetropia (Eye disorders) | 0 | 1
Lacrimation Increased (Eye disorders) | 8 | 4
Ocular Hyperaemia (Eye disorders) | 1 | 2
Optic Atrophy (Eye disorders) | 1 | 0
Papilloedema (Eye disorders) | 1 | 0
Periorbital Oedema (Eye disorders) | 1 | 1
Periorbital Swelling (Eye disorders) | 0 | 1
Photophobia (Eye disorders) | 6 | 2
Photopsia (Eye disorders) | 5 | 0
Vision Blurred (Eye disorders) | 17 | 12
Visual Field Defect (Eye disorders) | 2 | 1
Visual Impairment (Eye disorders) | 7 | 4
Vitreous Floaters (Eye disorders) | 1 | 3
Xerophthalmia (Eye disorders) | 0 | 1
Abdominal Distension (Gastrointestinal disorders) | 2 | 3
Abdominal Pain (Gastrointestinal disorders) | 10 | 7
Abdominal Pain Upper (Gastrointestinal disorders) | 11 | 7
Anal Incontinence (Gastrointestinal disorders) | 1 | 0
Aphthous Ulcer (Gastrointestinal disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 126 | 97
Dental Caries (Gastrointestinal disorders) | 1 | 1
Dental Paraesthesia (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 47 | 31
Dry Mouth (Gastrointestinal disorders) | 13 | 2
Dyspepsia (Gastrointestinal disorders) | 14 | 10
Dysphagia (Gastrointestinal disorders) | 5 | 2
Enterocolitis (Gastrointestinal disorders) | 1 | 0
Eructation (Gastrointestinal disorders) | 1 | 0
Flatulence (Gastrointestinal disorders) | 3 | 2
Gastritis (Gastrointestinal disorders) | 2 | 1
Gastrointestinal Inflammation (Gastrointestinal disorders) | 1 | 0
Gastrointestinal Pain (Gastrointestinal disorders) | 0 | 2
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 5 | 5
Gingival Bleeding (Gastrointestinal disorders) | 2 | 0
Gingival Pain (Gastrointestinal disorders) | 1 | 2
Haematemesis (Gastrointestinal disorders) | 2 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 3 | 4
Hyperaesthesia Teeth (Gastrointestinal disorders) | 1 | 0
Hypoaesthesia Oral (Gastrointestinal disorders) | 2 | 0
Impaired Gastric Emptying (Gastrointestinal disorders) | 1 | 0
Large Intestinal Stenosis (Gastrointestinal disorders) | 1 | 0
Lip Swelling (Gastrointestinal disorders) | 0 | 1
Mouth Haemorrhage (Gastrointestinal disorders) | 1 | 0
Mouth Ulceration (Gastrointestinal disorders) | 2 | 0
Nausea (Gastrointestinal disorders) | 205 | 122
Odynophagia (Gastrointestinal disorders) | 0 | 2
Oral Dysaesthesia (Gastrointestinal disorders) | 1 | 0
Oral Pain (Gastrointestinal disorders) | 1 | 1
Paraesthesia Oral (Gastrointestinal disorders) | 1 | 0
Proctalgia (Gastrointestinal disorders) | 0 | 1
Rectal Haemorrhage (Gastrointestinal disorders) | 2 | 1
Salivary Hypersecretion (Gastrointestinal disorders) | 1 | 0
Stomatitis (Gastrointestinal disorders) | 3 | 3
Toothache (Gastrointestinal disorders) | 2 | 3
Upper Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 158 | 53
Administration Site Dysaesthesia (General disorders) | 0 | 1
Asthenia (General disorders) | 33 | 28
Catheter Site Pain (General disorders) | 4 | 0
Catheter Site Thrombosis (General disorders) | 3 | 0
Chest Discomfort (General disorders) | 1 | 0
Chest Pain (General disorders) | 3 | 1
Chills (General disorders) | 6 | 4
Discomfort (General disorders) | 0 | 2
Disease Progression (General disorders) | 1 | 0
Face Oedema (General disorders) | 8 | 5
Fatigue (General disorders) | 188 | 170
Feeling Abnormal (General disorders) | 1 | 0
Feeling Cold (General disorders) | 2 | 0
Feeling Drunk (General disorders) | 1 | 0
Gait Disturbance (General disorders) | 72 | 15
General Physical Health Deterioration (General disorders) | 6 | 11
Generalised Oedema (General disorders) | 1 | 0
Granuloma (General disorders) | 0 | 1
Impaired Healing (General disorders) | 0 | 1
Induration (General disorders) | 0 | 1
Influenza Like Illness (General disorders) | 13 | 5
Infusion Site Discomfort (General disorders) | 1 | 0
Infusion Site Extravasation (General disorders) | 0 | 1
Infusion Site Irritation (General disorders) | 1 | 0
Infusion Site Pain (General disorders) | 8 | 0
Infusion Site Phlebitis (General disorders) | 2 | 0
Injection Site Bruising (General disorders) | 2 | 0
Injection Site Discomfort (General disorders) | 1 | 0
Injection Site Pain (General disorders) | 13 | 0
Injection Site Reaction (General disorders) | 9 | 0
Localised Oedema (General disorders) | 0 | 1
Malaise (General disorders) | 5 | 5
Mucosal Inflammation (General disorders) | 2 | 0
Non-Cardiac Chest Pain (General disorders) | 1 | 0
Oedema (General disorders) | 2 | 2
Oedema Peripheral (General disorders) | 18 | 8
Pain (General disorders) | 5 | 3
Peripheral Swelling (General disorders) | 2 | 0
Pyrexia (General disorders) | 34 | 11
Scar Inflammation (General disorders) | 0 | 2
Temperature Regulation Disorder (General disorders) | 1 | 0
Thirst (General disorders) | 1 | 0
Vascular Device Occlusion (General disorders) | 1 | 0
Vessel Puncture Site Pain (General disorders) | 1 | 0
Xerosis (General disorders) | 0 | 1
Cholestasis (Hepatobiliary disorders) | 0 | 1
Drug-Induced Liver Injury (Hepatobiliary disorders) | 1 | 0
Allergic Oedema (Immune system disorders) | 0 | 1
Drug Hypersensitivity (Immune system disorders) | 1 | 0
Hypersensitivity (Immune system disorders) | 1 | 1
Seasonal Allergy (Immune system disorders) | 1 | 0
Anal Abscess (Infections and infestations) | 1 | 0
Bacterial Infection (Infections and infestations) | 0 | 1
Brain Abscess (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 9 | 2
Bronchitis Viral (Infections and infestations) | 1 | 0
Candida Infection (Infections and infestations) | 6 | 3
Catheter Site Infection (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 2
Conjunctivitis (Infections and infestations) | 1 | 4
Conjunctivitis Viral (Infections and infestations) | 0 | 2
Covid-19 (Infections and infestations) | 1 | 1
Cystitis (Infections and infestations) | 4 | 2
Cytomegalovirus Infection (Infections and infestations) | 0 | 1
Device Related Infection (Infections and infestations) | 2 | 0
Device Related Sepsis (Infections and infestations) | 1 | 0
Ear Infection (Infections and infestations) | 1 | 0
Encephalomyelitis (Infections and infestations) | 1 | 0
Enterocolitis Infectious (Infections and infestations) | 1 | 0
Escherichia Urinary Tract Infection (Infections and infestations) | 0 | 1
Folliculitis (Infections and infestations) | 2 | 0
Fungal Infection (Infections and infestations) | 0 | 2
Gastroenteritis (Infections and infestations) | 4 | 3
Gastroenteritis Viral (Infections and infestations) | 2 | 0
Gingivitis (Infections and infestations) | 1 | 0
Hepatitis A (Infections and infestations) | 0 | 1
Herpes Dermatitis (Infections and infestations) | 1 | 0
Herpes Simplex (Infections and infestations) | 1 | 0
Herpes Simplex Reactivation (Infections and infestations) | 0 | 2
Herpes Virus Infection (Infections and infestations) | 0 | 1
Herpes Zoster (Infections and infestations) | 10 | 7
Herpes Zoster Infection Neurological (Infections and infestations) | 1 | 0
Infection (Infections and infestations) | 2 | 0
Influenza (Infections and infestations) | 1 | 4
Kidney Infection (Infections and infestations) | 1 | 0
Lower Respiratory Tract Infection (Infections and infestations) | 2 | 0
Meningitis Bacterial (Infections and infestations) | 1 | 1
Mucosal Infection (Infections and infestations) | 0 | 1
Nail Infection (Infections and infestations) | 1 | 0
Nasopharyngitis (Infections and infestations) | 7 | 3
Oral Candidiasis (Infections and infestations) | 6 | 6
Oral Fungal Infection (Infections and infestations) | 2 | 0
Oral Herpes (Infections and infestations) | 3 | 2
Oropharyngeal Candidiasis (Infections and infestations) | 0 | 1
Otitis Externa (Infections and infestations) | 1 | 0
Pharyngitis (Infections and infestations) | 2 | 1
Pneumocystis Jirovecii Pneumonia (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 7 | 4
Pneumonia Chlamydial (Infections and infestations) | 1 | 0
Postoperative Wound Infection (Infections and infestations) | 1 | 1
Rash Pustular (Infections and infestations) | 1 | 1
Respiratory Tract Infection (Infections and infestations) | 2 | 1
Respiratory Tract Infection Viral (Infections and infestations) | 1 | 0
Retinitis (Infections and infestations) | 0 | 1
Rhinitis (Infections and infestations) | 2 | 0
Sepsis (Infections and infestations) | 2 | 0
Septic Shock (Infections and infestations) | 1 | 0
Sinusitis (Infections and infestations) | 3 | 1
Skin Infection (Infections and infestations) | 1 | 0
Staphylococcal Bacteraemia (Infections and infestations) | 1 | 0
Subcutaneous Abscess (Infections and infestations) | 1 | 0
Subdural Abscess (Infections and infestations) | 1 | 0
Tooth Abscess (Infections and infestations) | 1 | 0
Tooth Infection (Infections and infestations) | 0 | 1
Tracheitis (Infections and infestations) | 1 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 7 | 7
Urinary Tract Infection (Infections and infestations) | 13 | 10
Urosepsis (Infections and infestations) | 1 | 0
Vestibular Neuronitis (Infections and infestations) | 1 | 0
Viral Rash (Infections and infestations) | 0 | 1
Wound Infection (Infections and infestations) | 1 | 0
Animal Bite (Injury, poisoning and procedural complications) | 1 | 0
Brain Herniation (Injury, poisoning and procedural complications) | 0 | 1
Chemical Phlebitis (Injury, poisoning and procedural complications) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 2 | 3
Eye Contusion (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 35 | 15
Femoral Neck Fracture (Injury, poisoning and procedural complications) | 0 | 1
Foot Fracture (Injury, poisoning and procedural complications) | 0 | 1
Foreign Body In Eye (Injury, poisoning and procedural complications) | 0 | 1
Head Injury (Injury, poisoning and procedural complications) | 2 | 0
Incision Site Dermatitis (Injury, poisoning and procedural complications) | 0 | 1
Incision Site Swelling (Injury, poisoning and procedural complications) | 1 | 0
Infusion Related Reaction (Injury, poisoning and procedural complications) | 13 | 0
Joint Injury (Injury, poisoning and procedural complications) | 0 | 1
Ligament Sprain (Injury, poisoning and procedural complications) | 1 | 1
Limb Injury (Injury, poisoning and procedural complications) | 0 | 1
Lumbar Vertebral Fracture (Injury, poisoning and procedural complications) | 2 | 1
Pneumocephalus (Injury, poisoning and procedural complications) | 0 | 1
Post Procedural Discomfort (Injury, poisoning and procedural complications) | 0 | 1
Procedural Pain (Injury, poisoning and procedural complications) | 2 | 0
Pseudomeningocele (Injury, poisoning and procedural complications) | 1 | 1
Radiation Alopecia (Injury, poisoning and procedural complications) | 1 | 3
Radiation Necrosis (Injury, poisoning and procedural complications) | 2 | 0
Radiation Skin Injury (Injury, poisoning and procedural complications) | 17 | 31
Radius Fracture (Injury, poisoning and procedural complications) | 0 | 1
Scar (Injury, poisoning and procedural complications) | 0 | 1
Skin Abrasion (Injury, poisoning and procedural complications) | 1 | 0
Skin Laceration (Injury, poisoning and procedural complications) | 0 | 2
Skin Wound (Injury, poisoning and procedural complications) | 1 | 0
Spinal Fracture (Injury, poisoning and procedural complications) | 1 | 0
Subdural Haematoma (Injury, poisoning and procedural complications) | 0 | 1
Tendon Rupture (Injury, poisoning and procedural complications) | 1 | 0
Thermal Burn (Injury, poisoning and procedural complications) | 1 | 1
Toxicity To Various Agents (Injury, poisoning and procedural complications) | 1 | 0
Vascular Access Site Haematoma (Injury, poisoning and procedural complications) | 1 | 0
Wound (Injury, poisoning and procedural complications) | 1 | 1
Wound Dehiscence (Injury, poisoning and procedural complications) | 0 | 1
Alanine Aminotransferase Increased (Injury, poisoning and procedural complications) | 18 | 12
Amylase Increased (Injury, poisoning and procedural complications) | 1 | 0
Aspartate Aminotransferase Increased (Injury, poisoning and procedural complications) | 8 | 4
Blood Alkaline Phosphatase Increased (Injury, poisoning and procedural complications) | 3 | 0
Blood Bilirubin Increased (Injury, poisoning and procedural complications) | 6 | 0
Blood Calcium Decreased (Injury, poisoning and procedural complications) | 1 | 0
Blood Cholesterol Increased (Injury, poisoning and procedural complications) | 0 | 2
Blood Creatinine (Injury, poisoning and procedural complications) | 1 | 0
Blood Creatinine Increased (Injury, poisoning and procedural complications) | 9 | 5
Blood Folate Decreased (Injury, poisoning and procedural complications) | 1 | 0
Blood Glucose Increased (Injury, poisoning and procedural complications) | 0 | 1
Blood Lactate Dehydrogenase Increased (Injury, poisoning and procedural complications) | 3 | 0
Blood Potassium Decreased (Injury, poisoning and procedural complications) | 2 | 0
Blood Sodium Decreased (Injury, poisoning and procedural complications) | 1 | 0
Blood Testosterone Decreased (Injury, poisoning and procedural complications) | 1 | 0
Blood Uric Acid Increased (Injury, poisoning and procedural complications) | 0 | 1
C-Reactive Protein Increased (Injury, poisoning and procedural complications) | 4 | 0
Cardiac Murmur (Injury, poisoning and procedural complications) | 1 | 0
Computerised Tomogram Head (Injury, poisoning and procedural complications) | 0 | 1
Electrocardiogram Qt Prolonged (Injury, poisoning and procedural complications) | 1 | 0
Gamma-Glutamyltransferase Increased (Injury, poisoning and procedural complications) | 8 | 4
Hepatic Enzyme Increased (Injury, poisoning and procedural complications) | 1 | 0
International Normalised Ratio Increased (Injury, poisoning and procedural complications) | 0 | 1
Lymphocyte Count Decreased (Injury, poisoning and procedural complications) | 15 | 17
Neutrophil Count Decreased (Injury, poisoning and procedural complications) | 11 | 15
Neutrophil Count Increased (Injury, poisoning and procedural complications) | 1 | 1
Oxygen Saturation Decreased (Injury, poisoning and procedural complications) | 1 | 0
Platelet Count Decreased (Injury, poisoning and procedural complications) | 25 | 37
Propionibacterium Test Positive (Injury, poisoning and procedural complications) | 1 | 0
Serum Ferritin Decreased (Injury, poisoning and procedural complications) | 0 | 1
Transaminases Increased (Injury, poisoning and procedural complications) | 3 | 0
Urine Output Increased (Injury, poisoning and procedural complications) | 0 | 1
Vitamin B12 Decreased (Injury, poisoning and procedural complications) | 0 | 1
Vitamin D Decreased (Injury, poisoning and procedural complications) | 0 | 1
Weight Decreased (Injury, poisoning and procedural complications) | 48 | 23
Weight Increased (Injury, poisoning and procedural complications) | 13 | 13
White Blood Cell Count (Injury, poisoning and procedural complications) | 0 | 1
White Blood Cell Count Decreased (Injury, poisoning and procedural complications) | 7 | 11
White Blood Cell Count Increased (Injury, poisoning and procedural complications) | 2 | 0
Decreased Appetite (Metabolism and nutrition disorders) | 64 | 52
Dehydration (Metabolism and nutrition disorders) | 10 | 0
Diabetes Mellitus (Metabolism and nutrition disorders) | 1 | 0
Dyslipidaemia (Metabolism and nutrition disorders) | 0 | 1
Glucose Tolerance Impaired (Metabolism and nutrition disorders) | 0 | 2
Gout (Metabolism and nutrition disorders) | 1 | 0
Hypercreatininaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 12 | 7
Hyperkalaemia (Metabolism and nutrition disorders) | 3 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 1 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 6 | 5
Hypomagnesaemia (Metabolism and nutrition disorders) | 3 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 3 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 2 | 0
Hypoproteinaemia (Metabolism and nutrition disorders) | 1 | 0
Increased Appetite (Metabolism and nutrition disorders) | 1 | 0
Lipomatosis (Metabolism and nutrition disorders) | 1 | 0
Obesity (Metabolism and nutrition disorders) | 0 | 1
Polydipsia (Metabolism and nutrition disorders) | 0 | 1
Steroid Diabetes (Metabolism and nutrition disorders) | 0 | 1
Type 2 Diabetes Mellitus (Metabolism and nutrition disorders) | 0 | 1
Vitamin B12 Deficiency (Metabolism and nutrition disorders) | 2 | 0
Vitamin D Deficiency (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 19 | 9
Back Pain (Musculoskeletal and connective tissue disorders) | 18 | 13
Bone Pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Extremity Contracture (Musculoskeletal and connective tissue disorders) | 0 | 1
Facial Asymmetry (Musculoskeletal and connective tissue disorders) | 3 | 1
Flank Pain (Musculoskeletal and connective tissue disorders) | 1 | 3
Joint Stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0
Joint Swelling (Musculoskeletal and connective tissue disorders) | 3 | 0
Limb Discomfort (Musculoskeletal and connective tissue disorders) | 1 | 0
Mastication Disorder (Musculoskeletal and connective tissue disorders) | 1 | 0
Mobility Decreased (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 7 | 4
Muscle Tightness (Musculoskeletal and connective tissue disorders) | 1 | 1
Muscle Twitching (Musculoskeletal and connective tissue disorders) | 2 | 1
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 31 | 21
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 3 | 1
Musculoskeletal Disorder (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 1 | 2
Musculoskeletal Stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 11 | 8
Myokymia (Musculoskeletal and connective tissue disorders) | 1 | 0
Myopathy (Musculoskeletal and connective tissue disorders) | 4 | 2
Neck Pain (Musculoskeletal and connective tissue disorders) | 11 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 2
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 7 | 5
Pain In Jaw (Musculoskeletal and connective tissue disorders) | 7 | 1
Sjogren's Syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0
Tendon Discomfort (Musculoskeletal and connective tissue disorders) | 0 | 1
Tendon Disorder (Musculoskeletal and connective tissue disorders) | 1 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Trismus (Musculoskeletal and connective tissue disorders) | 1 | 0
Brain Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Glioblastoma Multiforme (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Malignant Neoplasm Progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8 | 5
Melanocytic Naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases To Meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Neoplasm Progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Peritumoural Oedema (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Squamous Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Squamous Cell Carcinoma Of Skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Ageusia (Nervous system disorders) | 1 | 1
Agraphia (Nervous system disorders) | 0 | 1
Akathisia (Nervous system disorders) | 2 | 1
Alexia (Nervous system disorders) | 1 | 0
Amnesia (Nervous system disorders) | 9 | 4
Anosmia (Nervous system disorders) | 2 | 3
Aphasia (Nervous system disorders) | 48 | 22
Apraxia (Nervous system disorders) | 1 | 5
Ataxia (Nervous system disorders) | 70 | 2
Balance Disorder (Nervous system disorders) | 42 | 9
Brain Oedema (Nervous system disorders) | 14 | 11
Brain Stem Haematoma (Nervous system disorders) | 1 | 0
Cerebellar Syndrome (Nervous system disorders) | 1 | 0
Cerebral Cyst (Nervous system disorders) | 1 | 1
Cerebral Haemorrhage (Nervous system disorders) | 3 | 0
Cerebral Ischaemia (Nervous system disorders) | 1 | 0
Cerebral Venous Thrombosis (Nervous system disorders) | 1 | 0
Clonus (Nervous system disorders) | 0 | 1
Cognitive Disorder (Nervous system disorders) | 19 | 12
Complex Regional Pain Syndrome (Nervous system disorders) | 0 | 2
Coordination Abnormal (Nervous system disorders) | 4 | 1
Depressed Level Of Consciousness (Nervous system disorders) | 6 | 2
Disturbance In Attention (Nervous system disorders) | 19 | 7
Dizziness (Nervous system disorders) | 71 | 31
Dizziness Postural (Nervous system disorders) | 0 | 2
Dysaesthesia (Nervous system disorders) | 3 | 1
Dysarthria (Nervous system disorders) | 45 | 12
Dysgeusia (Nervous system disorders) | 16 | 26
Dysgraphia (Nervous system disorders) | 1 | 0
Dyskinesia (Nervous system disorders) | 0 | 2
Dyslexia (Nervous system disorders) | 1 | 0
Dyspraxia (Nervous system disorders) | 2 | 1
Encephalopathy (Nervous system disorders) | 3 | 1
Epilepsy (Nervous system disorders) | 6 | 6
Extensor Plantar Response (Nervous system disorders) | 1 | 0
Facial Paralysis (Nervous system disorders) | 2 | 0
Facial Paresis (Nervous system disorders) | 1 | 3
Fine Motor Skill Dysfunction (Nervous system disorders) | 1 | 0
Frontotemporal Dementia (Nervous system disorders) | 0 | 1
Generalised Tonic-Clonic Seizure (Nervous system disorders) | 2 | 2
Gerstmann's Syndrome (Nervous system disorders) | 0 | 1
Head Discomfort (Nervous system disorders) | 1 | 0
Head Titubation (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 163 | 92
Hemianopia (Nervous system disorders) | 0 | 3
Hemianopia Heteronymous (Nervous system disorders) | 0 | 1
Hemianopia Homonymous (Nervous system disorders) | 0 | 1
Hemiparaesthesia (Nervous system disorders) | 1 | 0
Hemiparesis (Nervous system disorders) | 23 | 17
Hydrocephalus (Nervous system disorders) | 2 | 3
Hypersomnia (Nervous system disorders) | 10 | 1
Hypertonia (Nervous system disorders) | 1 | 0
Hypoaesthesia (Nervous system disorders) | 10 | 5
Intracranial Pressure Increased (Nervous system disorders) | 4 | 2
Ischaemic Stroke (Nervous system disorders) | 1 | 0
Lethargy (Nervous system disorders) | 9 | 2
Leukoencephalopathy (Nervous system disorders) | 1 | 0
Loss Of Consciousness (Nervous system disorders) | 1 | 0
Memory Impairment (Nervous system disorders) | 19 | 19
Monoparesis (Nervous system disorders) | 4 | 0
Monoplegia (Nervous system disorders) | 1 | 0
Motor Dysfunction (Nervous system disorders) | 5 | 2
Movement Disorder (Nervous system disorders) | 1 | 0
Myoclonus (Nervous system disorders) | 1 | 0
Nervous System Disorder (Nervous system disorders) | 5 | 2
Neuralgia (Nervous system disorders) | 2 | 0
Neurologic Neglect Syndrome (Nervous system disorders) | 1 | 1
Neurological Decompensation (Nervous system disorders) | 5 | 2
Neurological Symptom (Nervous system disorders) | 1 | 0
Neuromyelitis Optica Spectrum Disorder (Nervous system disorders) | 1 | 0
Neuropathy Peripheral (Nervous system disorders) | 3 | 0
Nystagmus (Nervous system disorders) | 6 | 0
Optic Neuritis (Nervous system disorders) | 1 | 0
Paraesthesia (Nervous system disorders) | 13 | 6
Partial Seizures (Nervous system disorders) | 4 | 5
Peripheral Sensory Neuropathy (Nervous system disorders) | 4 | 3
Polyneuropathy (Nervous system disorders) | 0 | 1
Post Herpetic Neuralgia (Nervous system disorders) | 3 | 1
Postural Tremor (Nervous system disorders) | 1 | 0
Presyncope (Nervous system disorders) | 2 | 1
Psychomotor Hyperactivity (Nervous system disorders) | 2 | 0
Pyramidal Tract Syndrome (Nervous system disorders) | 0 | 1
Quadrantanopia (Nervous system disorders) | 1 | 1
Radicular Pain (Nervous system disorders) | 1 | 0
Resting Tremor (Nervous system disorders) | 1 | 0
Restless Legs Syndrome (Nervous system disorders) | 2 | 0
Sciatic Nerve Neuropathy (Nervous system disorders) | 1 | 0
Seizure (Nervous system disorders) | 35 | 38
Sensory Disturbance (Nervous system disorders) | 1 | 0
Slow Speech (Nervous system disorders) | 2 | 0
Somnolence (Nervous system disorders) | 17 | 3
Speech Disorder (Nervous system disorders) | 10 | 2
Spinal Cord Oedema (Nervous system disorders) | 1 | 0
Status Epilepticus (Nervous system disorders) | 1 | 1
Subdural Effusion (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 2 | 5
Taste Disorder (Nervous system disorders) | 3 | 2
Temporal Lobe Epilepsy (Nervous system disorders) | 1 | 1
Tension Headache (Nervous system disorders) | 1 | 1
Tongue Biting (Nervous system disorders) | 1 | 0
Tonic Clonic Movements (Nervous system disorders) | 0 | 1
Tremor (Nervous system disorders) | 19 | 13
Trigeminal Neuralgia (Nervous system disorders) | 0 | 1
Tunnel Vision (Nervous system disorders) | 1 | 0
Upper Motor Neurone Lesion (Nervous system disorders) | 0 | 1
Vasogenic Cerebral Oedema (Nervous system disorders) | 3 | 4
Visual Field Defect (Nervous system disorders) | 3 | 0
Abnormal Dreams (Psychiatric disorders) | 7 | 0
Abulia (Psychiatric disorders) | 1 | 2
Adjustment Disorder (Psychiatric disorders) | 1 | 0
Affect Lability (Psychiatric disorders) | 3 | 1
Affective Disorder (Psychiatric disorders) | 1 | 0
Agitation (Psychiatric disorders) | 17 | 4
Alcohol Abuse (Psychiatric disorders) | 0 | 1
Anhedonia (Psychiatric disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 33 | 18
Apathy (Psychiatric disorders) | 1 | 0
Attention Deficit Hyperactivity Disorder (Psychiatric disorders) | 1 | 1
Bradyphrenia (Psychiatric disorders) | 3 | 2
Confusional State (Psychiatric disorders) | 62 | 24
Deja Vu (Psychiatric disorders) | 1 | 0
Delirium (Psychiatric disorders) | 11 | 2
Delusion (Psychiatric disorders) | 2 | 0
Depressed Mood (Psychiatric disorders) | 7 | 1
Depression (Psychiatric disorders) | 19 | 14
Depressive Symptom (Psychiatric disorders) | 0 | 1
Derealisation (Psychiatric disorders) | 1 | 0
Discouragement (Psychiatric disorders) | 1 | 0
Disorientation (Psychiatric disorders) | 3 | 2
Euphoric Mood (Psychiatric disorders) | 0 | 1
Hallucination (Psychiatric disorders) | 115 | 1
Hallucination, Auditory (Psychiatric disorders) | 4 | 0
Hallucination, Visual (Psychiatric disorders) | 20 | 1
Hallucinations, Mixed (Psychiatric disorders) | 3 | 0
Illusion (Psychiatric disorders) | 1 | 0
Impulsive Behaviour (Psychiatric disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 87 | 36
Irritability (Psychiatric disorders) | 5 | 2
Libido Decreased (Psychiatric disorders) | 1 | 1
Logorrhoea (Psychiatric disorders) | 1 | 0
Mania (Psychiatric disorders) | 4 | 0
Mental Fatigue (Psychiatric disorders) | 1 | 0
Mental Status Changes (Psychiatric disorders) | 0 | 1
Nervousness (Psychiatric disorders) | 4 | 1
Nightmare (Psychiatric disorders) | 14 | 1
Obsessive Thoughts (Psychiatric disorders) | 1 | 0
Panic Attack (Psychiatric disorders) | 1 | 1
Paranoia (Psychiatric disorders) | 3 | 0
Perseveration (Psychiatric disorders) | 2 | 0
Personality Change (Psychiatric disorders) | 5 | 1
Phobia (Psychiatric disorders) | 1 | 0
Procedural Anxiety (Psychiatric disorders) | 0 | 1
Psychomotor Retardation (Psychiatric disorders) | 3 | 0
Psychotic Disorder (Psychiatric disorders) | 1 | 0
Reading Disorder (Psychiatric disorders) | 1 | 0
Restlessness (Psychiatric disorders) | 1 | 2
Sleep Disorder (Psychiatric disorders) | 8 | 0
Acute Kidney Injury (Renal and urinary disorders) | 1 | 0
Azotaemia (Renal and urinary disorders) | 1 | 0
Chromaturia (Renal and urinary disorders) | 1 | 0
Cystitis Noninfective (Renal and urinary disorders) | 0 | 1
Dysuria (Renal and urinary disorders) | 1 | 1
Haematuria (Renal and urinary disorders) | 2 | 3
Incontinence (Renal and urinary disorders) | 1 | 0
Micturition Urgency (Renal and urinary disorders) | 3 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 2
Nocturia (Renal and urinary disorders) | 1 | 2
Pollakiuria (Renal and urinary disorders) | 2 | 4
Polyuria (Renal and urinary disorders) | 1 | 2
Proteinuria (Renal and urinary disorders) | 2 | 0
Renal Failure (Renal and urinary disorders) | 2 | 0
Urethral Intrinsic Sphincter Deficiency (Renal and urinary disorders) | 1 | 0
Urge Incontinence (Renal and urinary disorders) | 0 | 1
Urinary Incontinence (Renal and urinary disorders) | 8 | 3
Amenorrhoea (Reproductive system and breast disorders) | 0 | 1
Balanoposthitis (Reproductive system and breast disorders) | 1 | 0
Benign Prostatic Hyperplasia (Reproductive system and breast disorders) | 1 | 0
Breast Inflammation (Reproductive system and breast disorders) | 1 | 0
Erectile Dysfunction (Reproductive system and breast disorders) | 1 | 1
Heavy Menstrual Bleeding (Reproductive system and breast disorders) | 0 | 1
Pelvic Pain (Reproductive system and breast disorders) | 1 | 1
Prostatic Pain (Reproductive system and breast disorders) | 1 | 0
Pruritus Genital (Reproductive system and breast disorders) | 0 | 1
Vaginal Discharge (Reproductive system and breast disorders) | 1 | 0
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 29 | 15
Dry Throat (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 8 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 9 | 15
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 | 4
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 7 | 4
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonia Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 1
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 5 | 4
Respiratory Tract Congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rhinitis Allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Sinus Congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Sleep Apnoea Syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Upper-Airway Cough Syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Acne (Skin and subcutaneous tissue disorders) | 0 | 2
Alopecia (Skin and subcutaneous tissue disorders) | 73 | 99
Cold Sweat (Skin and subcutaneous tissue disorders) | 1 | 0
Decubitus Ulcer (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 8 | 10
Dermatitis Acneiform (Skin and subcutaneous tissue disorders) | 2 | 3
Dermatitis Allergic (Skin and subcutaneous tissue disorders) | 0 | 2
Dermatitis Bullous (Skin and subcutaneous tissue disorders) | 0 | 1
Dermatitis Contact (Skin and subcutaneous tissue disorders) | 0 | 2
Drug Eruption (Skin and subcutaneous tissue disorders) | 0 | 1
Dry Skin (Skin and subcutaneous tissue disorders) | 8 | 8
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 | 1
Eczema (Skin and subcutaneous tissue disorders) | 3 | 1
Erythema (Skin and subcutaneous tissue disorders) | 9 | 7
Erythema Multiforme (Skin and subcutaneous tissue disorders) | 1 | 0
Hirsutism (Skin and subcutaneous tissue disorders) | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0
Intertrigo (Skin and subcutaneous tissue disorders) | 1 | 0
Miliaria (Skin and subcutaneous tissue disorders) | 1 | 0
Nail Bed Inflammation (Skin and subcutaneous tissue disorders) | 0 | 1
Night Sweats (Skin and subcutaneous tissue disorders) | 1 | 0
Onycholysis (Skin and subcutaneous tissue disorders) | 1 | 0
Pain Of Skin (Skin and subcutaneous tissue disorders) | 1 | 4
Petechiae (Skin and subcutaneous tissue disorders) | 1 | 4
Photosensitivity Reaction (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 18 | 13
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 2
Purpura (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 18 | 4
Rash Erythematous (Skin and subcutaneous tissue disorders) | 1 | 0
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 7 | 4
Rash Pruritic (Skin and subcutaneous tissue disorders) | 1 | 1
Scar Pain (Skin and subcutaneous tissue disorders) | 3 | 2
Sensitive Skin (Skin and subcutaneous tissue disorders) | 1 | 1
Skin Disorder (Skin and subcutaneous tissue disorders) | 0 | 1
Skin Exfoliation (Skin and subcutaneous tissue disorders) | 1 | 0
Skin Irritation (Skin and subcutaneous tissue disorders) | 2 | 0
Skin Lesion (Skin and subcutaneous tissue disorders) | 1 | 0
Skin Striae (Skin and subcutaneous tissue disorders) | 0 | 1
Skin Toxicity (Skin and subcutaneous tissue disorders) | 2 | 0
Skin Ulcer (Skin and subcutaneous tissue disorders) | 1 | 0
Stevens-Johnson Syndrome (Skin and subcutaneous tissue disorders) | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 4 | 1
Deep Vein Thrombosis (Vascular disorders) | 8 | 3
Embolism (Vascular disorders) | 2 | 0
Flushing (Vascular disorders) | 4 | 1
Haematoma (Vascular disorders) | 2 | 2
Hot Flush (Vascular disorders) | 5 | 2
Hypertension (Vascular disorders) | 14 | 9
Hypotension (Vascular disorders) | 5 | 2
Jugular Vein Thrombosis (Vascular disorders) | 1 | 0
Lymphoedema (Vascular disorders) | 1 | 0
Orthostatic Hypotension (Vascular disorders) | 0 | 1
Peripheral Ischaemia (Vascular disorders) | 0 | 1
Phlebitis (Vascular disorders) | 7 | 0
Raynaud's Phenomenon (Vascular disorders) | 1 | 0
Subclavian Vein Thrombosis (Vascular disorders) | 1 | 0
Thrombophlebitis (Vascular disorders) | 6 | 0
Thrombophlebitis Superficial (Vascular disorders) | 5 | 0
Thrombosis (Vascular disorders) | 0 | 2
Varicose Ulceration (Vascular disorders) | 1 | 0
Vascular Pain (Vascular disorders) | 2 | 0
Venous Thrombosis (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-06-20): https://cdn.clinicaltrials.gov/large-docs/95/NCT03345095/Prot_000.pdf
  • Statistical Analysis Plan (2021-03-18): https://cdn.clinicaltrials.gov/large-docs/95/NCT03345095/SAP_001.pdf